CLINICAL TRIAL: NCT06507124
Title: Qualitative Thematic Analysis of Non-radiologist Clinicians' Approach to CT Body Interpretation
Brief Title: Rapid Examination of Acute CT
Acronym: REACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Lancashire Hospitals NHS Trust (Other)
Collaborators: University of Central Lancashire (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 336924
Record Dates: First submitted 2024-03-01; First posted 2024-07-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Behavior
Keywords: Computed tomography; Medical education
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Doctors of various grades will be Invited to take part in the study. Thematic analysis will be used to assess the recordings.
Masking Description: The identify of the participant will not be known to the analysis team
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm (Experimental)
  Interventions: Other: This is observational with no intervention

INTERVENTIONS:
Other: This is observational with no intervention — This is observational with no intervention

SUMMARY:
CT scans are becoming increasingly prevalent in medicine. These are reviewed by radiologists and formal report provided. A recent survey suggests that non-radiologists are increasingly being expected to be able to interpret pathology on CT scans, however there is limited training provided in medical school and specialty training schemes.

This study aims to qualitatively analyse how non-radiologists of different seniority and specialties approach CT body scan interpretation. This will be done by recording participants as they look at a pre-selected CT scan.

The data will be reviewed with a thematic analysis. The eventual aim is to develop a CT interpretation system, which can be used by the non-radiologist to look for important pathology on a CT scan of the body

DETAILED DESCRIPTION:
A recent survey published in a local conference (Master 2023) asked 100 junior doctors across 16 Trusts in the UK (including ELHT and MFT) about their experience of CT. This showed that confidence in CT requesting and interpretation is very limited. From the same survey it seems that CT is very superficially taught in medical schools with no system given for interpretation. 90% of those surveyed said they would benefit from more educational resources in CT. The investigators hope to develop a CT interpretation resource to help the non-radiologist when looking at CT scans. This study aims to see how non-radiologists currently approach a CT scan to gain understanding of the needs of the new resources.

There is no similar study in the literature investigating how the non-radiologist approaches CT scans. There has been investigation of foundation doctors experience in radiology, however the focus was on plain xrays, not CT interpretation.

The investigators plan to use a thematic analysis in data interpretation. Rationale for using Thematic analysis.

* Recognised method of identifying patterns/ themes in qualitative data for learning and teaching research.
* Provides a flexible methodology approach which is not reliant on a particular educational theory. Hence it is able to deal with relatively uncharted area of how non-radiologists interpret radiological images.

Process of thematic analysis . Using the 6-step approach. Step Aims Comments

1. Data familiarisation Studying the transcripts & video with notes on initial impressions.
2. Initial codes derived Grouping data in a meaningful and systematic way.
3. Search for themes Discerning any significant pattern in the data.
4. Review themes Review the support for each theme and if they cover the entire data set.
5. Define themes Clear description of each theme covering the points it is addressing, any sub-themes it contains and how they relate to one-another.
6. Write-up Report on the key points, from this study, which are influencing CT scan interpretation and how it could be taught.

   * The proposed study is using an inductive and latent level approach for the data analysis. This was selected as it allows the flexibility to look beyond what is being said. The semantic approach was considered too restrictive as it assumes a predefined understanding of the subjects' cognitive strategy in dealing with image interpretation. In contrast, by combining the oral presentation with the manipulation of the image and the answering of key questions there will be a better chance of appreciating the underlying cognitive approach being employed.
   * Open coding will be used for the transcripts analysed so far. This allows them to be modified under the influence of more data.
   * Currently,qualitative data analytic software (e.g. ATLAS, Nvivo etc.) are not using.

The reason being the researcher's need for first-hand familiarisation with a novel dataset. Once this preliminary phase has been carried out consideration will be given to using UCLan's access to Nvivo. This decision will take into account personal preferences, experiences with the preliminary data and the anticipated size of the data base.

• Once preliminary themes have been proposed a review will be made to see which codes they address. Unlinked codes will prompt further analysis of the themes, considered of new themes or development of sub-themes. This iterative process continues with new data until a steady state is achieved and no new themes are being generated.

ELIGIBILITY:
Inclusion Criteria:

* Doctors will be recruited from East Lancashire Hospitals NHS Trust (ELHT) and Participant Identification Centre (PIC) sites via a convenience sampling method.
* Participants must be currently working in UK NHS acute specialties (ED, Medicine, Surgery, etc).
* Includes doctor grades from Foundation to Consultant. Senior radiology trainees and consultants will also be recruited as an expert comparison.

Exclusion Criteria:

* Non-clinical doctors
* Radiologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
Observe the difference in CT interpretation technique between traditionally trained radiology consultants and other clinicians of varying seniorities | 1 year
  Process of thematic analysis. The proposed study is using an inductive and latent level approach for the data analysis. This was selected as it allows the flexibility to look beyond what is being said. By combining the oral presentation with the manipulation of the image and the answering of key questions we feel there will be a better chance of appreciating the underlying cognitive approach being employed.
  Open coding will be used for the transcript analysis. This allows them to be modified under the influence of more data.
  Once preliminary themes have been proposed a review will be made to see which codes they address. Unlinked codes will prompt further analysis of the themes, considered of new themes or development of sub-themes. This iterative process continues with new data until a steady state is achieved and no new themes are being generated.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua J Lauder, MBChB FRCR, Principal Investigator — ELHT
Locations (1):
- East Lancashire Hospitals NHS Trust, Blackburn, United Kingdom

IPD SHARING:
Plan to Share IPD: No